CLINICAL TRIAL: NCT00614601
Title: A Phase II Study of Low Dose Algenpantucel-L (HyperAcute Pancreas) Cancer Vaccine in Subjects With Surgically Resected Pancreatic Cancer
Brief Title: Low Dose Vaccine Study for Surgically Resected Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor proceeded with a phase III study for same indication.
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG0305; OBA#0704-844
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; vaccine therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vaccine + chemo + chemoradiation therapy
  Interventions: Biological: HyperAcute(R)-Pancreatic Cancer Vaccine
- 2 (Experimental): Vaccine Only
  Interventions: Biological: HyperAcute(R)-Pancreatic Cancer Vaccine

INTERVENTIONS:
Biological: HyperAcute(R)-Pancreatic Cancer Vaccine — 100 million vaccine cells will be injected intradermally for up to 14 vaccinations over approximately 8 months
  Other Names: HAPa-1 and HAPa-2 vaccine components

SUMMARY:
To assess the response for subjects with pancreatic cancer that have undergone surgical resection and treatment with a vaccine given with or without chemotherapy and chemoradiation.

DETAILED DESCRIPTION:
Unfortunately, despite the best clinical efforts and breakthroughs in biotechnology, most patients diagnosed with pancreatic cancer continue to die from their disease in a very short period of time. The primary reason for this is the short progression time of the disease; in fact, most patients with pancreatic cancer have symptoms at the time of the diagnosis. Moreover, lack of any single agent or procedure to have any significant impact on long term survival rates further contributes to poor prognostic outcomes observed with this disease.

These reasons are the major causes of cancer progression that are usually discussed when considering treatment options for patients with disease that continues to grow and spread. However, another important part of the body should be considered-- the immune system. Scientists have clearly shown that pancreatic cancer cells as well as other cancer cells produce a number of abnormal proteins or abnormal amounts of certain proteins not found in normal cells. Normally one would expect a patient to develop an immune response against these abnormal proteins found in their cancer and attack them much the way we would fight off an infection from a foreign bacteria or virus. However, for reasons that scientists do not fully understand, the immune system fails to respond to these abnormal proteins and does not attack the cancer cells. This human clinical trial proposes a new way to make the immune system recognize the cancer and encourage it to attack the cancer cells.

Many people are familiar with the idea of transplants between people of organs like the kidneys or heart. When an organ transplant between two people is completed one of the problems that can occur is rejection of the donated organ by the recipient. This can occur because the immune system of the patient who receives the organ attacks the donated organ. If you were to attempt to transplant a pig heart to a human the rejection would be dramatically stronger than when organs are transplanted between two people. This is partly because lower animals express sugar-protein patterns on the surface of their cells that humans do not. In fact, our immune systems can quickly recognize tissues from lower mammals such as the pig or the mouse and destroys them.

In this project, we propose to put a mouse gene into human pancreatic cancer cells that produces these abnormal sugar patterns and stimulates the immune system to attack the pancreatic cancer. This strategy works well to kill other human cancer cells in the laboratory, but it needs to be tried in pancreatic cancer patients to see if it will be effective. We propose to test this new treatment in patients with pancreatic cancer who have undergone tumor resection to see if it can stop or slow recurrence of tumors in these patients. Patients will be injected with an anti-tumor vaccine consisting of a mixture of two types of dead human pancreatic cancer cells that have been genetically altered to express the mouse gene responsible for making this abnormal sugar-protein on the cells.

ELIGIBILITY:
Inclusion Criteria:

* A histological diagnosis of adenocarcinoma of the pancreas. The patient's pathology must be reviewed and confirmed by the clinical site's Pathology Department.
* AJCC Stage I or II Pancreatic carcinoma. Patients must have undergone surgical resection for the tumor and extent of resection must be either R0 (complete resection with grossly and microscopically negative margins or resection) or R1 (grossly negative but positive microscopically margins of resection).
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Serum albumin ≥ 2.0 gm/dL.
* Expected survival ≥ 6 months.
* Subjects must have a negative serology for HIV prior to entering study.
* Subjects must be able to take in ≥ 1500 calories daily.
* Adequate organ function including:
* Marrow: WBC ≥3000/mm3 and platelets ≥100,000/mm3.
* Hepatic: serum total bilirubin ≤ 2 x ULN mg/dL, ALT (SGPT) and AST (SGOT) ≤3 x upper limit of normal (ULN).
* Renal: serum creatinine (sCr) ≤2.0 x ULN, or creatinine clearance (Ccr) ≥30 mL/min.
* First vaccination must be within 6 weeks after surgery.
* Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able give written informed consent to participate.
* All subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product, and for one month after the last immunization.

Exclusion Criteria:

* Age <18-years-old.
* Active metastases.
* Other malignancy within five years, unless the probability of recurrence of the prior malignancy is <5%. Patient's curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant.
* Current, active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subjects taking chronic systemic corticosteroid therapy for any reason are not eligible. Subjects may receive steroids as prophylactic anti-emetics, not to exceed 10 mg Decadron weekly. Subjects may also receive pulse doses for Gemcitabine hypersensitivity, not to exceed Decadron 8 mg BID x 3 days prior to start day of Gemcitabine. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require chronic systemic corticosteroids after beginning vaccination, will be removed from study.
* Significant or uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias within the last six months.
* Active infection or antibiotics within 1-week prior to study, including unexplained fever (temp > 38.1C).
* Autoimmune disease (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), etc.). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis) or a serious illness in medical opinion of the clinical investigator.
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.).
* A known allergy to any component of the vaccine or cell lines.
* Pregnant or nursing women due to the unknown effects of vaccination on the developing fetus or newborn infant. (For patients with child bearing potential, a βHCG must be completed within 7 days of first vaccination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this Phase II trial is to assess disease-free survival (DFS) at one (1) year following initiation of treatment as the primary endpoint of the study in subjects treated with the HyperAcute®-Pancreatic Cancer Vaccine | One year

SECONDARY OUTCOMES:
We will use overall survival and adverse events rates as secondary endpoints. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Charles J. Link, M.D., Study Chair — NewLink Genetics Corporation
Locations (1):
- University of Louisville, Louisville, Kentucky, United States